CLINICAL TRIAL: NCT05765006
Title: A Phase I Dose-escalation Study Evaluate the Safety Tolerability Pharmacokinetics(PK) and Pharmacodynamics(PD) of Relma-cel in Subjects With Moderate to Severe Active Systemic Lupus Erythematosus (SLE)
Brief Title: CD19-CART(Relma-cel) for Moderate to Severe Active Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029012
Record Dates: First submitted 2023-02-06; First posted 2023-03-13 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Relma-cel; Systemic lupus erythematosus; CD19-CART
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relma-cel be administrated in four dose level (Experimental)
  Interventions: Biological: Relma-cel

INTERVENTIONS:
Biological: Relma-cel — CD19-targeted Chimeric AntigenReceptor (CAR) T Cells; Relma-cel be administrated at four dose level:25×106 CAR+ T cells、50×106 CAR+ T cells、100×106 CAR+ T cells/150×106 CAR+ T cells

SUMMARY:
This is a phase I, open-label, single-arm, multicenter study to asess the safety tolerability pharmacokinetics and pharmacodynamics of Relma-cel in moderate or severe active systemic lupus erythematosus (SLE) subjects in China.

DETAILED DESCRIPTION:
This is a phase I, open-label, single-arm, multicenter study to asess the safety tolerability pharmacokinetics(PK) and pharmacodynamics(PD) of Relma-cel in moderate or severe active systemic lupus erythematosus (SLE) subjects in China.

There will be 4 dose level (15x106 CAR+ T cells as the back up dose ,25x106 CAR+ T cells as the starting dose 、50x106 CAR+ T cells and 100x106(or 150 x106CAR+ T cells）Dose escalation, to evaluate the safety、 tolerability of Relma-cel in adult subjects of SLE and determine RP2D .

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form (ICF) voluntarily.
2. At the time of signing the ICF, you must be between 18 and 70 years old (inclusive), male or female.
3. A diagnosis of SLE according to the 1997 revised criteria of the American College of Rheumatology (ACR).
4. The history of SLE prior to screening was at least 6 months, and the disease remained active at least 2 months after the use of a stable standard SLE regimen prior to screening.

Standard treatment regimen refers to the steady use of any of the following (alone or in combination) : corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and other immunosuppressants or immunomodulators including azathioprine, Mycophenolate Mofetil, cyclophosphamide, methotrexate, leflunomide, tacrolimus, and cyclosporine.

Oral corticosteroids must meet the following requirements:

1. Prednisone (or equivalent) ≥7.5 mg/ day, and ≤30 mg/ day.
2. There is no minimum daily dose requirement for corticosteroids when used in combination with immunosuppressants.
3. At least 8 weeks of treatment prior to screening, and the dose must be kept stable for > 2 weeks.

5. Screening is positive for antinuclear antibodies, and/or anti-DS-DNA antibodies, and/or anti-Smith antibodies.

6. SELENA-SLEDAI score ≥8 during the screening period. Score ≥6 for SELENA-SLEDAI clinical symptoms (except for low complement and/or anti-DS-DNA antibodies) if low complement and/or anti-DS-DNA antibody score is present.

Exclusion Criteria:

1. Severe lupus nephritis (defined as proteinuria > 6 g/24h or serum creatinine > 2.5 mg/dL or 221 μmol/L), treatment with active nephritis with Prohibited drugs, hemodialysis, or prednisone ≥100 within 8 weeks prior to screening mg/d or equivalent glucocorticoid therapy ≥14 days.
2. Prior to screening, other lupus crises, such as active central nervous system lupus, severe hemolytic anemia, severe thrombocytopenic purpura, severe agranulocytosis, severe myocardial damage, severe lupus pneumonia or pulmonary hemorrhage, severe lupus hepatitis, and severe vasculitis.
3. Clinically significant central nervous system diseases or pathological changes not caused by lupus prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
4. Combined with other autoimmune diseases, systematic treatment is needed.
5. History of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
6. IgA deficiency was present during screening (serum IgA level < 10 mg/dL)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT rate | 3 months
  The incidence of dose-limiting toxicity
determine RP2D | 3 months
  To determine RP2D(Phase 2 recommended dose)

SECONDARY OUTCOMES:
SELENA-SLEDAI （Safety of Estrogens in Systemic Lupus Erythematosus National Assessment） score； 0 to 4 is basically no disease activity; 5 to 9 is light activity; 10 to 14 is moderate activity;≥15 is considered heavy activity. | 3 months
  SELENA-SLEDAI score taken up to 3 months after CD19 cCAR T cells infusion
BILAG -2004（updated version of british isles lupus assessment group ） level；The BILAG 2004 index categorizes disease activity into 5 different levels from A-E.Grade A represents very active disease. | 3 months
  BILAG-2004 level taken up to 3 months after CD19 cCAR T cells infusion
PGA (physician global assessment) score,The PGA scale ranges from "no disease activity" (0) to the "most severe disease activity" (3).the score is between 0 to 3. | 3 months
  PGA score taken up to 3 months after CD19 cCAR T cells infusion
Autoantibody detection | 3 months
  Autoantibody detection up to 3 months after CD19 cCAR T cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: yu Hu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; liangjing Lv, Principal Investigator — Renji Hospital Shanghai Jiaotong University School of Medical
Locations (1):
- Relma-cel Medical, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaufman JL, Deak ST, Erdman W. Radionuclide scans to define patterns of occult myonecrosis. N J Med. 1986 Feb;83(2):101-3. No abstract available. PMID 3005930
- [Derived] Shu J, Xie W, Mei C, Ren A, Ke S, Ma M, Zhou Z, Hu Y, Mei H. Safety and clinical efficacy of Relmacabtagene autoleucel (relma-cel) for systemic lupus erythematosus: a phase 1 open-label clinical trial. EClinicalMedicine. 2025 Apr 30;83:103229. doi: 10.1016/j.eclinm.2025.103229. eCollection 2025 May. PMID 40386685